CLINICAL TRIAL: NCT02124616
Title: National Registry for Egyptian Pediatric Neuromuscular Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sahar M.A. Hassanein, MD, Professor of Pediatrics, Ain Shams University
Other Study IDs: EGYPT PED-NMD 2014
Record Dates: First submitted 2014-04-25; First posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Spinal Muscular Atrophy; Muscular Dystrophy; Muscle Diseases; Myasthenic Syndromes; Polyneuropathies
Keywords: spinal muscular atrophy; Muscular dystrophy; Muscle diseases; myasthenic syndromes; Polyneuropathies; Myopathies
MeSH Terms: conditions — Muscular Atrophy, Spinal; Muscular Dystrophies; Lambert-Eaton Myasthenic Syndrome; Polyneuropathies; Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Neuromuscular diseases: Prospective cohort of children with inherited or acquired neuromuscular diseases.

SUMMARY:
Our aim is to establish multi-center national Egyptian database of information for inherited and acquired neuromuscular diseases in infants and children from 0 to 18 years of age.

DETAILED DESCRIPTION:
Aims: An open-ended multi-center, national Egyptian study to collect and analyze data for children with Neuromuscular Diseases (NMD) inherited NMD (spinal muscular atrophy (SMA), Duchenne/Becker and congenital muscular dystrophies (DMD/BMD, CMD), congenital myopathies, and congenital myasthenic syndromes) and acquired NMD (neuropathies, myasthenia gravis and myositis).

Participants: Eligible infants and children with inherited and acquired neuromuscular diseases.

DESIGN: This study is a prospective cohort study.

Outcome measures: Motor development assessment, respiratory and cardiac examination.

ELIGIBILITY:
Inclusion Criteria:

* Weakness, hypotonia.
* Nerve conduction study and electromyographic confirmation of lower motor neuron affection.

Exclusion Criteria:

* Chromosomal diseases.
* Malformations and deformations.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children from birth to 18 years of age with inherited or acquired neuromuscular diseases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Functional motor ability | 1 year
  Motor power in acquired acute neuromuscular diseases will be assessed at admission and morbidity and mortality at discharge from hospital.
  Functional motor ability will be performed every 3 months for children with inherited neuromuscular diseases.

SECONDARY OUTCOMES:
Cardio-pulmonary function | 12 months
  Pulmonary and cardiac function impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar MA Hassanein, MD, PhD, Study Chair — Pediatric Department, Children's Hospital, Faculty of Medicine, Ain Shams University
Locations (1):
- Pediatric Department, Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Abassia, Egypt

REFERENCES:
- See also: Faculty of Medicine, Ain Shams University website — http://med.asu.edu.eg/
- See also: Ain Shams University web site — http://www.asu.edu.eg/